CLINICAL TRIAL: NCT06531148
Title: A Clinical and Microbiological Assessment of the Efficacy of Chemo-mechanical Caries Removal Versus Conventional Caries Removal Methods in Children: Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0303023PP
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-10

CONDITIONS: Chemo-Mechanical Caries Removal

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled clinical trial with split-mouth technique
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemo-mechanical caries removal (Experimental): A Chemo-mechanical caries removal agent for one side of the bilateral carious teeth (selected randomly). Application of the material will be done according to the manufacturer's instructions
  Interventions: Other: Chemo-mechanical caries removal
- Conventional drilling method (Other): * In this group, caries removal was performed using a low-speed handpiece with a carbon steel round bur.
  * The cavities were then examined using the same criteria that had been used with Group I to assess for any remaining caries.
  * After caries removal, a dentin sample was taken from the cavity floor in both groups using a sterile sharp spoon excavator.
  * The dentin sample was transported to a sterile screw-cap vial for bacterial count examination.
  Interventions: Other: Chemo-mechanical caries removal

INTERVENTIONS:
Other: Chemo-mechanical caries removal — Chemo-mechanical were be used as a Chemo-mechanical caries removal agent for one side of the bilateral carious teeth (selected randomly). Application of the material were be done according to the manufacturer's instructions (20). The material will be applied with a blunt spoon excavator and left for 2 minutes allowing the chemistry to work. The decayed dentin which becomes soft (due to the action of the material) was being scraped away using a blunt excavator in a pendulum movement without pressure. If necessary, the procedure will be repeated to get healthy dentin. The cavity will be visually inspected by caries detector dye to assess the complete removal of the carious dentin.

SUMMARY:
This study will be conducted to Assess the clinical and microbiological efficacy of chemomechanical caries removal (CarieMove® Gel) versus conventional excavation method in children.

The assessed parameters will be:

* Efficacy of caries removal.
* Pain reaction and mean time required for the treatment.
* Total bacterial count before and after treatment.

DETAILED DESCRIPTION:
Subjects:

A total of 30 children 7-9 years old with no history of systematic disease will be recruited from the out-patient pediatric dental clinic, Faculty of Dentistry, Mansoura University.

Each child with the following criteria will be eligible for the present study (22).

Inclusion criteria:

1. Cooperative child
2. Each child has two bilateral first permanent molars with simple Class 1 occlusal caries involving dentin.
3. The carious first permanent molars are free from clinical and radiographic evidence of pulp involvement.
4. The selected molars should have normal structure and morphology.

Exclusion criteria:

1. Un-cooperative child
2. Molars with clinical and radiographic signs of pulp involvement.
3. Children with special health care needs.
4. Molars which have already been restored or have developmental anomaly.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative child
2. Each child has two bilateral first permanent molars with simple Class 1 occlusal caries involving dentin.
3. The carious first permanent molars are free from clinical and radiographic evidence of pulp involvement.
4. The selected molars should have normal structure and morphology.

Exclusion Criteria:

* 1- Un-cooperative child 2- Molars with clinical and radiographic signs of pulp involvement. 3- Children with special health care needs. 4- Molars which have already been restored or have developmental anomaly.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2024-10-02 (Estimated); Study Completion 2024-11-11 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | 11.2 ± 3.3 min
  A-Efficacy:
  B- Child satisfaction and pain experience:
  C-Time assessment

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Dentistry, Al Mansurah, El-dahlewa
  - Dentistry, Al Mansurah